CLINICAL TRIAL: NCT02329808
Title: Clinical Validation of a Dried Blood Spot (DBS) Method for the Analysis of Immunosuppressive and Antifungal Drugs in Pediatric Patients (Part of the PROTECT Study).
Brief Title: Clinical Validation of a Dried Blood Spot Method for Analysis of Immunosuppressives and Antifungals in Pediatrics
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF 14.02
Record Dates: First submitted 2014-12-19; First posted 2015-01-01 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hematologic Diseases; Oncology Problem; Kidney Diseases; Transplantation Infection
Keywords: TDM; dried blood spot; immunosuppressive; antifungal
MeSH Terms: conditions — Hematologic Diseases; Kidney Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma without DNA, blood with DNA and dried blood spot (with DNA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- Mycophenolic acid: Patients treated for their regular patient care with mycophenolic acid.
  Interventions: Procedure: blood drawing
- Cyclosporin: Patients treated for their regular patient care with cyclosporin.
  Interventions: Procedure: blood drawing
- Tacrolimus: Patients treated for their regular patient care with tacrolimus.
  Interventions: Procedure: blood drawing
- Sirolimus: Patients treated for their regular patient care with sirolimus.
  Interventions: Procedure: blood drawing
- Everolimus: Patients treated for their regular patient care with everolimus.
  Interventions: Procedure: blood drawing
- Voriconazole: Patients treated for their regular patient care with voriconazole.
  Interventions: Procedure: blood drawing
- Posaconazole: Patients treated for their regular patient care with posaconazole.
  Interventions: Procedure: blood drawing
- Itraconazole+metabolite: Patients treated for their regular patient care with itraconazole.
  Interventions: Procedure: blood drawing
- Fluconazole: Patients treated for their regular patient care with fluconazole.
  Interventions: Procedure: blood drawing

INTERVENTIONS:
Procedure: blood drawing — The association between conventional venous sampling and finger prick dried blood spot (DBS) will be associated by drawing blood in both ways.

SUMMARY:
This is a clincial validation study of a dried blood spot (DBS) method for the analysis of immunosuppressive and antifungal agents currently subject of therapeutic drug monitoring (TDM) in a pediatric population.

The primary goal is to clinically validate a finger prick DBS method compared to conventional venous sampling for the analysis of 5 immunosuppressive and 4 azole antifungal drugs in the pediatric population. Secondairy goals include feasibility of the finger prick DBS method in the target population, to design an inventory of costs that will be incurred in future health-economic analyses and to construct a population PK model based on the available data collected for the primariy goal.

DETAILED DESCRIPTION:
Therapeutic drug monitoring (TDM) offers the possibility to individualize and improve a patient's pharmacological treatment, based on the measurement of drug concentrations in biological samples. Conventionally, TDM is performed with blood or plasma obtained by venous blood sampling. This method is associated with several challenges such as i) the need for the patient to travel to the hospital or health center; ii) special conditions for sample transport to guarantee stability of the analyte and to decrease the biohazard risk; iii) sampling times not always representing the preferable peak or trough concentrations; iv) the method being invasive and v) delay of the outcome of the analyses with regard to the outpatient visit.

The Dried Blood Spot (DBS) may offer a solution for all these challenges. DBS is thought to offer benefits over plasma venous sampling for TDM. The main purpose of the PROTECT (Personalized treatment of immunosuppressive and antifungal drugs through continuous home based monitoring with Dried Blood Spot sampling techniques in pediatric patients) study is to improve therapeutic management and patient participation in pediatric patients treated with antifungal and immunosuppressive agents. PROTECT is mainly financed by a ZonMW grant 'Goed Gebruik Geneesmiddelen'.

Four patient organizations are actively involved in the PROTECT study.

Objective of the study:

Primairy To clinically validate a finger prick DBS method compared to conventional venous sampling for the analysis of 5 immunosuppressive and 4 azole antifungal drugs in the pediatric population. Secondairy

* Feasibility of the novel finger prick DBS method in the pediatric population will be assessed. This includes scoring of relevant characteristics (attributes) of blood drawing methods for TDM, evaluation of the experience and attitude of both patients and parents regarding finger prick DBS sampling and evaluation of the understanding of the written instructions provided for performing the finger prick at home. The data obtained in this validation study will be used for the implementation of the DBS in therapeutic drug monitoring (TDM) being a less invasive procedure, and as a base for a discrete choice-experiment as part of the HTA.
* To design an inventory of types of costs that will be incurred in the process of DBS-based and conventional TDM as a preparation step for later health economic analysis.
* Data from this study will be used to construct a population pharmacokinetic model to optimize dosing and design new guidelines.

This is an observational mono-centre study in which DBS sampling is compared with conventional sampling for TDM in a steady state situation.

Clearly, information on feasibility of DBS sampling in children and on costs relevant to DBS sampling in children can only be obtained through actual sampling in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 2 and 18 years
* Admitted to the Radboudumc pediatric ward
* Having a venous catheter
* Treated with at least 1 of the 9 drugs of interest
* The drug concentration being at steady state
* Signed informed consent

Exclusion Criteria:

* Parents and/or patients are not able to understand the Dutch language

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric hemato-oncology and primariy immunodeficient patients and pediatric renal transplantation patients.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
drug concentration | predose, 2 samples postdose, max 6 hours post dose
  The outcome measure is a composite of several blood concentrations, obtained by three individual blood drawing moments per patient. The related endpoint is the evaluation of the association between the concentration obtained by venous sampling and the concentration obtained by means of DBS sampling. The predictive performance of the DBS method as a measure for the venous concentration will be evaluated.

SECONDARY OUTCOMES:
Questionnaire | 1 day
  The related endpoint is the response to a questionnaire. Results will be used to prepare implementation of the novel method for home-based monitoring as well as to prepare a HTA analysis.
costs | 2 years
  Costs of blood drawing methods will be collected.The cost types will function as a basis for future HTA analysis of this novel sampling method compared to conventional venous sampling.
Area under the curve | 6h period
  Blood concentrations will be used to calculate the area under the concentration time curve (AUC). The outcome measure will be a composite of population estimates of the pharmacokinetic parameters AUC, maximal concentration (Cmax), time to maximal concentration (Tmax), clearance (CL), volume of distribution (Vd) and elimination half-life (t1/2).

CONTACTS AND LOCATIONS:
Overall Officials: Roger Bruggemann, PharmD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No